CLINICAL TRIAL: NCT00983593
Title: A Randomized Clinical Study of a Mind-Body Approach to Domestic Violence Offender Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 34135
Record Dates: First submitted 2009-08-25; First posted 2009-09-24 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Domestic Violence; Intimate Partner Violence
Keywords: Mind Body Bridging; Domestic Violence Offender Treatment; Batterer Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Group Therapy (Experimental): Group therapy following the Mind-Body Bridging program.
  Interventions: Behavioral: Mind-Body Bridging

INTERVENTIONS:
Behavioral: Mind-Body Bridging — 16 weeks of weekly Mind-Body Bridging group treatment lasting 60-90 minutes per session.

SUMMARY:
The focus of the present study is to examine the relative efficacy of a mind-body method, know as Mind-Body Bridging, of treating DV offenders as compared to a "treatment as usual" (TAU) approach. The study will be conducted on-site at ACES, a non-profit agency that provides licensed domestic violence offender and substance abuse treatment services in the Salt Lake City area.

DETAILED DESCRIPTION:
Mind-Body Bridging Program (MBBP) was developed by Stanley Block, M.D. over the last decade drawing from his more than 30 years of experience in clinical psychiatry and awareness training. In his book Come To Your Senses: Demystifying the Mind-Body Connection (Block & Block, 2005, 2007), he demonstrates how people can regulate their emotions through "bridging", a technique that brings one back to the present moment to experience and recognize thoughts, emotions and physical sensations. Bridging aims to reduce the impact of negative thought patterns that facilitate stress in the body. Bridging allows individuals to reconnect with a mind-body state that inherently relaxes and restores healthy natural functioning. MBBP is built on awareness practices that enable individuals to investigate their mental states at deeper levels for the purpose of calming their minds and relaxing their bodies. This can lead to reductions in activation of the stress system (stress is consistently implicated in the progression of many mental and physical diseases), with the prospect of potentially alleviating many detrimental health conditions. According to Block & Block (2005, 2007), the critical source of ill-being in humans is rooted in the "Identity System" (IS), which is composed of self-centered thoughts, beliefs and emotions. The IS emphasizes separation, incompleteness, and self-interest, creating an identity that lacks authenticity. In essence, the IS interferes with one's natural functioning in everyday life by effectively cutting one off from one's natural self-healing abilities, and this typically results in constricting and closing down the present-moment awareness that is provided by one's senses. MBBP teaches how using bridging techniques, one can identify and "rest" the IS with its associated negativity and bodily tension, thereby creating more opportunities for improving quality of life and for functioning more naturally.

ELIGIBILITY:
Inclusion Criteria:

* Court ordered to completed domestic violence offender treatment

Exclusion Criteria:

* Do not speak English

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Official Recidivism | 12-18 months

SECONDARY OUTCOMES:
Quality of Life Measure- Form-36 (SF-36) | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- ACES, Salt Lake City, Utah, United States